CLINICAL TRIAL: NCT05432297
Title: Preventive Randomized Study Regarding Physical Activity Intervention for Patients Receiving Radiotherapy for Head and Neck Cancer: the Effect of Preventive Intervention for Physical Activity, Function and Quality of Life
Brief Title: Preventive Physical Activity Intervention in Head and Neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lisa Tuomi, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2022-04-12; First posted 2022-06-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Neoplasms; Physical Inactivity
MeSH Terms: conditions — Head and Neck Neoplasms; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical exercise intervention (Experimental): The physical activity intervention is based on national guidelines of physical activity in cancer rehabilitation. A physiotherapist together with each patient will develop individual adaptations to the exercise protocol, with suggestions on which type of exercise the participant is able to perform depending on their daily condition. Suggestions on physical activity for good, bad and in-between-days will be listed in collaboration with the participant, and the participant will report number of minutes/day in each of the 3 physical activity levels stated.
  Interventions: Behavioral: Preventive physical exercise
- Control (No Intervention): The control group will receive general advice on the importance of physical activity during oncologic treatment, according to local clinical standard.

INTERVENTIONS:
Behavioral: Preventive physical exercise — Daily physical activity depending on daily condition
  Arms: Physical exercise intervention

SUMMARY:
The study includes patients with tumors of the oropharynx, larynx and hypopharynx scheduled to receive radiotherapy with curative intent (+/- chemotherapy). The patients will be randomized into either an intervention group (performing a preventive physical activity protocol before and during radiotherapy) or a control group not performing a specified physical exercise protocol. All patients will be in contact with with a speech language pathologist or a physical therapist weekly during radiotherapy. The study is expected to improve physical function and quality of life during and after oncologic treatment

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer (tumors of the oropharynx, pharynx, hypopharynx and larynx)
* Receiving radiohterapy (+/- chemotherapy) with curative intent

Exclusion Criteria:

* Surgery due to head and neck cancer
* Previous treatment for head and neck cancer
* Tracheostomized patients
* Inability to perform exercise intervention
* Inability to perform part of 6-minute walking test
* Inability to independently fill out questionnaires in Swedish
* Previous neurologic or neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Objectively measured physical activity | Up to 12 months
  Measured with an accelerometer. Measures time spent in different activities i minutes/day.
Subjectively measured physical activity - Saltin-Grimby | Up to 12 months
  Measured with the Saltin-Grimby physical activity level scale and the International Physical Activity Questionnaire.
Subjectively measured physical activity (IPAQ) | Up to 12 months
  Measured with the International Physical Activity Questionnaire

SECONDARY OUTCOMES:
Health related quality of life (HRQL) using the EORTC QLQ-C30 | Up to 5 years post radiotherapy
  Measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) core questionnaire (c30). Consists of 30 items divided into six functional domains (Physical, Role, Cognitive, Emotional, and Social Functioning and Global Quality of life), three symptom scales (Fatigue, Pain, and Nausea/Vomiting) and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). All domains range from 0-100. For the functional domains a higher score indicates good function, while for all other domains a high score indicates a high prevalence of symtoms, i.e. worse HRQL.
Health related quality of life (HRQL) using the EORTC QLQ H&N35 | Up to 5 years post radiotherapy
  Measured with the EORTC QLQ Head and neck module (HN35). It consists of 35 questions regarding symptoms more specific to the head and neck cancer population, and domain scores range from 0-100, where a higher score represents the prevalence of more symtoms, i.e. worse HRQL.
Trismus and jaw related symptoms | Up to 5 years post radiotherapy
  Patient Reported Outcomes (PRO) measured with Gothenburg Trismus Questionnaire (GTQ). The GTQ consists of 21 items divided into 3 domains; Jaw related problems, Eating limitations and Muscular tension and eight single items concerning facial pain, limitations in mouth opening and inabilities to function on social and working contexts. The GTQ domains range from 0-100 where 0 equals to absence of symtoms and 100 equals worst possible symptoms.
Dysphagia related symtoms | Up to 5 years post radiotherapy
  PRO measured with M.D Anderson Dysphagia Inventory (MDADI). This is a cancer-specific instrument measuring dysphagia, social function and quality of life in head and neck cancer patients. It consists of 19 items in four domains; emotional, physical, functional and global quality of life. The range for each subscale is 20-100 where 100 indicates best possible swallowing, i.e. better outcome.
Maximal Interincisal opening (MIO) | Up to 5 years post radiotherapy
  Jaw opening measured in millimeters
Body composition | Up to 12 months post radiotherapy
  Bioelectric impedance analysis.
Grip strength | Up to 12 months post radiotherapy
  Measured with the a hand dynamometer
6-minute walking test | Up to 12 months post radiotherapy
  Measures total walking distance during 6 minutes.

OTHER OUTCOMES:
Cost | Up to 5 years post radiotherapy
  The cost of intervention compared to usual care. Costs in Swedish crowns (SEK) for the intervention and all visits to healthcare during 5 years will be recorded.
Quality of life for cost-effectiveness analysis | Up to 5 years post radiotherapy
  The outcomes of intervention compared to usual care using European Quality of life 5 dimensions (EQ5D).
Quality Adjusted Life Years (QALY) | Up to 5 years post radiotherapy
  QALY is a measurement that combines health-related quality of life (HRQL) and life expectancy in one index. The index range between 0 and 1, where 0 equals death and 1 represents perfect health. Thus, 1 QALY corresponds to 1 year of perfect health. This is calculated using the EQ-5D.
Incremental Cost Effectiveness Ratio (ICER) | Up to 5 years post radiotherapy
  Incremental cost for each QALY for the intervention group will be calculated using a Markov model which combines the costs and EQ-5D. The ICER will then be compared to the maximum willingness to pay level which is SEK 500,000 (€55,000) according to the Swedish National Board of Health and Welfare.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tuomi, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden